CLINICAL TRIAL: NCT05212480
Title: Evaluation of the Efficacy and Safety of Zinc in Viral Infections
Acronym: VIZIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIZIR.COV
Record Dates: First submitted 2022-01-07; First posted 2022-01-28 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: After initial medical evaluation, every patient who meet the inclusion criteria, will receive randomly either Zinc or Placebo as detailed above according to the predetermined randomization. Patients enrolled in the zinc group received 25 mg of zinc twice a day for 15 days. Patients enrolled in the placebo group received 1 capsule twice a day for 15 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc arm (Active Comparator): patients received a pill containing 25 mg of zinc twice a day for 15 days
  Interventions: Dietary Supplement: Placebo
- Placebo (Placebo Comparator): patients received identical shape, smell, taste and color pill like the protocol treatment twice a day for 15 days
  Interventions: Dietary Supplement: Zinc

INTERVENTIONS:
Dietary Supplement: Zinc — For each patient included, a prescription regimen of zinc (in bisglycinate form) is proposed at a dose of 25 mgtwice a day for 15 days for the intervention arm. This dose of zinc is to be taken away from meals.
  Arms: Placebo
Dietary Supplement: Placebo — For each patient included, a prescription of an identical to the intervention arm concerning shape, smell, taste and color pill of placebo . This dose of zinc is to be taken away from meals.
  Arms: Zinc arm

SUMMARY:
The main objective of the clinical study is to evaluate the efficacy of Zinc supplementation in non-critically ill Covid-19 patients..

DETAILED DESCRIPTION:
The VIZIR study is a national, longitudinal, multi-centre study conducted over a 3-month follow-up period.

The priori hypothesis was that supplementation with zinc would reduce 30-day mortality and need to intensive care unit (ICU) admission among non critically ill patients with Covid-19.

The VIZIR study will be carried out in Tunisia at the level of consultations of general practitioners of both sectors : public and liberal, as well as in the emergency services of Monastir and Sousse.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over .
* Sars-Cov2 infection Diagnosed with RT PCR , Rapid Test or Chest CT-Scan performed within the less than 5 days of symptoms.

Exclusion Criteria:

* Patients who received zinc before the start of the protocol.
* heart, liver, malignancies, or renal failure (estimated glomerular filtration rate ≤30 mL/min/1.73 m2);
* Mental disorders .
* Chronic Dialysis.
* Hospitalisation in ICU (use of respiratory or cardiovascular organ support (oxygen delivered by high-flow nasal cannula, noninvasive or invasive mechanical ventilation, or the use of vasopressors or inotropes). .
* Known hypersensitivity to zinc.
* unsuitability for oral administration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Mortality rate. | 30 days
  death rate
need for ICU admission | 30 days
  Number of participants admitted to the Intensive care unit (ICU)
Combined_outcome | 30 days
  Death and/ or need for admission to the ICU for COVID-19 related complications.
treatment safety | 30 days
  rate of adverse events

SECONDARY OUTCOMES:
Need for hospitalization for patients followed up at home | 30 days
  Need for hospitalization for patients followed up initially at home
lenghth of stay in Hospital | 30 days
  days spent at hospital for patients followed up initially at home
resolution of COVID-19 symptoms | 30 days
  Time to resolution of COVID-19 symptoms [ Evaluated at day 15 and day 30 precising the Time at which the patient is completely symptom free and severity of symptoms .
need for oxygen therapy | 30 days
  Number of participants who needed oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nouira A semir, Pr, Principal Investigator — emergency department of Fattouma Bourguiba Monastir
Locations (1):
- EPS Fattouma Bourguiba Monastir, Monastir, Tunisia

REFERENCES:
- [Derived] Ben Abdallah S, Mhalla Y, Trabelsi I, Sekma A, Youssef R, Bel Haj Ali K, Ben Soltane H, Yacoubi H, Msolli MA, Stambouli N, Beltaief K, Grissa MH, Khrouf M, Mezgar Z, Loussaief C, Bouida W, Razgallah R, Hezbri K, Belguith A, Belkacem N, Dridi Z, Boubaker H, Boukef R, Nouira S. Twice-Daily Oral Zinc in the Treatment of Patients With Coronavirus Disease 2019: A Randomized Double-Blind Controlled Trial. Clin Infect Dis. 2023 Jan 13;76(2):185-191. doi: 10.1093/cid/ciac807. PMID 36367144